CLINICAL TRIAL: NCT04001660
Title: Subbrow Blepharoplasty Combined With Double Eyelid Surgery for Upper Eyelid Rejuvenation in Asian Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20192048-F-2
Record Dates: First submitted 2019-06-24; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-01

CONDITIONS: Subbrow Blepharoplasty;Double Eyelid Surgery； Orbicularis Oculi Muscle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subbrow Blepharoplasty Combined with Double Eyelid Surgery (Experimental): An upper incision is made along the inferior margin of the eyebrow. A lower incision is determined according to necessary amount of skin excision. Then the skin and subcutaneous tissue were excised. The orbicularis oculi muscle (OOM) was separated and an OOM flap dissection was extended to the width of 15mm. A dissected OOM flap was lifted up and three transverse 3-0 nylon sutures were placed to fix it to the periosteum and then covered by the upper myocutaneous flap of the supraorbital rim. Through eyelid-crease approach the supratarsal upper eyelid skin and orbital fat was excised, adjusted and reshaped double-fold eyelids at the same time.
  Interventions: Procedure: Subbrow Blepharoplasty Combined with Double Eyelid Surgery

INTERVENTIONS:
Procedure: Subbrow Blepharoplasty Combined with Double Eyelid Surgery — An upper incision is made along the inferior margin of the eyebrow. A lower incision is determined according to necessary amount of skin excision. Then the skin and subcutaneous tissue were excised. The orbicularis oculi muscle (OOM) was separated and an OOM flap dissection was extended to the width of 15mm. A dissected OOM flap was lifted up and three transverse 3-0 nylon sutures were placed to fix it to the periosteum and then covered by the upper myocutaneous flap of the supraorbital rim. Through eyelid-crease approach the supratarsal upper eyelid skin and orbital fat was excised, adjusted and reshaped double-fold eyelids at the same time.

SUMMARY:
Subbrow blepharoplasty combined with double eyelid surgery excising the subbrow skin and the supratarsal upper eyelid skin, lifting and fixing the OOM flap, meanwhile restoring the natural and symmetrical appearance, is a safe, effective, and durable way for treating patients presenting with dermatochalasis.

ELIGIBILITY:
Inclusion Criteria:

* Visual, lacrimal gland and eyelid functions were normal The eyes and eyebrows are aged between 35 and 65 years Informed consent was signed and approved by ethics review

Exclusion Criteria:

* Congenital craniofacial deformity, acquired craniofacial injury Scar constitution, pregnancy Mental illness

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) scores | postoperative 6month
  1, poor; 2, fair; 3, good; 4, very good; and 5, excellent

CONTACTS AND LOCATIONS:
Locations (1):
- Baoqiang Song, Xi'an, Shaanxi, China